CLINICAL TRIAL: NCT03565224
Title: Prospective Follow-up Study of CeSPACE XP - Titanium Coated PEEK Cages - for the Treatment of Degenerative Cervical Disc Disease
Brief Title: Study of Titanium-Coated PEEK Cages for Degenerative Disc Disease
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1702
Record Dates: First submitted 2018-05-25; First posted 2018-06-21 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Spinal Fusion; Cervical Vertebral Fusion
Keywords: Cervical vertebrae; Postoperative complications; Radiography; Spinal fusion; Coating
MeSH Terms: conditions — Klippel-Feil Syndrome; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cespace: The patients have been operated with Cespace Titanium Coated PEEK Cage for Degenerative Disc Disease between 2014 and 2017. All patients are invited to the Hospital for Follow-Up. Depending on the date of Initial Intervention the timeframe of follow-up for the individual Patient is 1 to 4 years.

SUMMARY:
Prospective Follow-up study of CeSPACE XP coated PEEK cages for the treatment of degenerative cervical disc disease

DETAILED DESCRIPTION:
Anterior cervical discectomy and fusion (ACDF) has been accepted as the standard procedure for the treatment of myelopathy and radiculopathy in the cervical spine. A tricortical iliac crest bone graft is the traditional inter-body fusion material that can show perfect bony fusion and maintain the patency of the neuroforamen. However, donor site complications were reported in fusion with an iliac bone graft, such as subcutaneous hematomas, infections, and chronic wound pain.

Currently, the titanium cage and polyetheretherketone (PEEK) cage are the two most common cages in clinical practice. The ideal cage should lead to a high fusion rate and prevent complications, such as subsidence and loss of correction.

Even though a titanium cage can provide long-term stabilization, increase lordosis, and increase foramina height compared with the iliac bone graft, some inferior clinical outcomes appeared in clinical practice. Loss of correction is a major complication of subsidence that may eventually affect cervical spinal function after the operation.

A modulus of elasticity close to cortical bone might contribute to advantages in stress distribution and load sharing, which can contribute to a lower subsidence rate and, thus, better clinical results, making PEEK cages more welcomed by surgeons.

It is supposed, that in the cervical fusion procedure, a porous coating of a PEEK cage will lead to favourable results. Therefore, the present study intends to show these results, in a larger patient cohort who received such a coated cervical cage.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who received a CeSPACE XP cage between August 2013 and January 2017

Exclusion Criteria:

* Pregnancy
* Patient consent not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) during Follow-Up | Once between 1 to 4 years postoperative
  The Neck Disability Index(NDI) is a modification of the Oswestry Low Back Pain Disability Index . It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain. The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. All the points can be summed to a total score.

SECONDARY OUTCOMES:
Patient Satisfaction at Follow-Up | Once between 1 to 4 years postoperative
  Patient self-reported satisfaction measured by a four-level scale: excellent, good, not satisfied, bad
Neck Pain at Follow-Up | Once between 1 to 4 years postoperative
  Patient self-reported Neck Pain measured by Visual Analogue Scale (VAS). The VAS is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Arm Pain during Follow-Up | Once between 1 to 4 years postoperative
  Patient self-reported Arm Pain measured by Visual Analogue Scale (VAS). The VAS is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Neurological Outcome at Follow-Up | 1 to 4 years follow-up
  Current neurological assessment at follow-up, measured by a four-level scale: no deficit, sensory deficit, motor deficit, sensory & motor deficit
Work Status at Follow-Up | Once between 1 to 4 years postoperative
  current profession and working level
Radiographic Evaluation of Mobility at Follow-Up | Once between 1 to 4 years postoperative
  Radiological evaluation: Fusion criteria 1: Degree of Flexion, Degree of Extension, Mobility (Extension-Flexion)
Radiographic Evaluation of Bone Bridges at Follow-Up | Once between 1 to 4 years postoperative
  Radiological evaluation: Fusion criteria 2: no bone bridges between adjacent vertebral bodies, Radiological densities visible compared to directly postop state, Bone Bridges linking adjacent vertebral bodies (anterior / posterior)
Radiographic Evaluation of Radiolucencies at Follow-Up | Once between 1 to 4 years postoperative
  Radiological evaluation: Fusion criteria 3: no radiolucent line along the implant end plate (0%), mild / under 25% radiolucencies, moderate / 25-50% radiolucencies, severe / more than 50% radiolucencies

OTHER OUTCOMES:
Rate of Patients with Adverse Events and Serious Adverse Events during Follow-up | Up to 4 years postoperative
  Number of Patients who had potential reoperations and revisions

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Arregui, Dr., MD, Principal Investigator — Hospital MAZ Zaragoza
Locations (1):
- Hospital MAZ Zaragoza, Zaragoza, Spain